CLINICAL TRIAL: NCT00017836
Title: Mechanisms Linking Depression to Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Viola Vaccarino MD/PhD, Professor And Chair, Emory University
Other Study IDs: IRB00024823; R01HL068630 (NIH); 970 (Other: NIH ID)
Record Dates: First submitted 2001-06-15; First posted 2001-06-15 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Depression; Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Depression; Cardiovascular Diseases; Heart Diseases

SUMMARY:
To examine the role of depression on risk for cardiovascular disease in twins.

DETAILED DESCRIPTION:
BACKGROUND:

Multiple studies have demonstrated a higher risk of cardiovascular disease and worse cardiovascular disease (CVD) prognosis associated with depression that appear to synergistically and significantly adversely impact health. Because these initial studies are observational, much work remains to understand this area. If these conditions are mechanistically inter-related, identification of both conditions in the same subject may provide a means of enhancing risk stratification and most appropriately targeting therapy. If the interaction between the conditions is causal not simply associative, appropriate therapy interventions can be designed and tested.

DESIGN NARRATIVE:

The project is designed to clarify the role of depression on CVD risk by using a co-twin study design. The study will examine twin pairs from the Vietnam Era Twin Registry (VET). Twin pairs will be invited to participate if they meet two criteria: (1) neither has a history of CVD as of 1990 and (2) one twin is diagnosed with depression as of 1992. The study investigates the effects of depression on two indicators of "early" CVD: coronary flow reserve, assessed by means of Positron Emission Tomography (PET) myocardial infusion imaging; and heart rate variability (HRV) assessed by ambulatory electrocardiographic monitoring. It is hypothesized that within each pair, the twins who have clinical depression will exhibit lower coronary vascular reserve and lower heart rate variability compared with their co-twins without a history of depression. Moreover, by comparing the size of the intra-pair difference in these parameters between depression discordant monozygotic and dizygotic twins an estimate of the relative contributions of gene and environmental factors can be ascertained. In addition to the PET and HRV assessments, subjects will complete the Statistical Clinical Interview of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV SCID) to document a history of depression, a psychometric battery including the Early Trauma Inventory and Hamilton Depression Scale, and such risk factors as cigarette smoking, physical activity, blood pressure and blood lipids, glucose and insulin, indices of inflammation and thrombogenicity including levels of reactive protein C, fibrinogen, and P-selectin, and neurohormones such as adrenocorticotropic hormone, cortisol, and dehydroepiandrosterone sulphate.

ELIGIBILITY:
No eligibility criteria

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viola Vaccarino — Emory University

REFERENCES:
- [Derived] Eufinger SC, Votaw J, Faber T, Ziegler TR, Goldberg J, Bremner JD, Vaccarino V. Habitual dietary sodium intake is inversely associated with coronary flow reserve in middle-aged male twins. Am J Clin Nutr. 2012 Mar;95(3):572-9. doi: 10.3945/ajcn.111.018077. Epub 2012 Jan 18. PMID 22258268
- [Derived] Karohl C, Su S, Kumari M, Tangpricha V, Veledar E, Vaccarino V, Raggi P. Heritability and seasonal variability of vitamin D concentrations in male twins. Am J Clin Nutr. 2010 Dec;92(6):1393-8. doi: 10.3945/ajcn.2010.30176. Epub 2010 Oct 13. PMID 20943799
- [Derived] Dai J, Ziegler TR, Bostick RM, Manatunga AK, Jones DP, Goldberg J, Miller A, Vogt G, Wilson PW, Jones L, Shallenberger L, Vaccarino V. High habitual dietary alpha-linolenic acid intake is associated with decreased plasma soluble interleukin-6 receptor concentrations in male twins. Am J Clin Nutr. 2010 Jul;92(1):177-85. doi: 10.3945/ajcn.2010.29305. Epub 2010 May 12. PMID 20463041